CLINICAL TRIAL: NCT03536403
Title: Study of Spino-pelvic Sagittal Balance by Vicon® Optoelectronic System - Model of Non-invasive Kyphosis
Brief Title: Study of Spino-pelvic Sagittal Balance by Vicon® Optoelectronic System
Acronym: VICON-SPINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016/066/HP
Record Dates: First submitted 2018-04-26; First posted 2018-05-24 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental): EOS X-rays is done with et without a kyphosis induced corset and 8-meters walk test measured by optoelectronic Vicon system with et without a kyphosis induced corset
  Interventions: Radiation: EOS X-rays; Other: 8-meters walk test

INTERVENTIONS:
Radiation: EOS X-rays — EOS X-rays is done with et without a kyphosis induced corset
Other: 8-meters walk test — 8-meters walk test measured by optoelectronic Vicon system with et without a kyphosis induced corset

SUMMARY:
Spinal diseases often induce gait disorders with multifactorial origins such as lumbar pain, radicular pain, neurologic complications, or spinal deformities. However, radiography does not permit an analysis of spinal dynamics; therefore, sagittal balance dynamics during gait remain largely unexplored. This prospective and controlled study try to assess the Vicon system for detecting sagittal spinopelvic imbalance and to determine the modification induced by ant induced anterior sagittal imbalance on the kinetics walking parameters

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Aged between 20 to 40 years
* Height between 165 to 190 centimeters
* Asymptomatic subjects from spinal point of view
* BMI < 30 kg/m²
* Affiliated to French Social Security
* Subjects having read the information note and signed informed consent

Exclusion Criteria:

* Subjects with neurological, vestibular, rheumatological or orthopedic pathology which can influence walking and balance
* Subjects with known spinal pathology
* Subjects with visible morphologic spinal deformity
* Subjects with significant visual impairment (visual acuity < 6/10) despite an optical correction port
* Subjects unable to walk without help
* Person placed under the safeguard of justice, guardianship or curatorship
* Subjects involved in other biomedical research during this study
* Subjects presenting an asymptomatic spinal pathology discovered at the inclusion on the spinal EOS images.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Variations in spino-pelvic sagittal balance measured by EOS X-ray | 1 hour
  Variations in spino-pelvic sagittal balances measured with et without a kyphosis induced corset measured by the GSC7 on EOS X-rays and by the C7-T10-Sacrum angle on optoelectronic Vicon system.

SECONDARY OUTCOMES:
Position of the ground point projection of the center of mass | 1 hour
  Position of the ground point projection of the center of mass with and without corset
vertical deceleration of the center of mass during the second part of the oscillating phase | 1 hour
  vertical deceleration of the center of mass during the second part of the oscillating phase with and without corset.
Velocity of the center of mass during the second part of the oscillating phase | 1 hour
  Velocity of the center of mass during the second part of the oscillating phase with and without corset.

CONTACTS AND LOCATIONS:
Overall Officials: Mourad OULD SLIMANE, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France